CLINICAL TRIAL: NCT03856476
Title: Early Markers of Endothelial and Renal Dysfunction in Children With Dyslipidemia
Brief Title: The Effect of Childhood Dyslipidemia on Endothelial and Renal Function
Status: Completed | Type: Observational
Sponsor: University of Ioannina (Other)
Collaborators: University Hospital, Ioannina (Other)
Responsible Party: Principal Investigator, Chrysoula Kosmeri, Principal Investigator, University of Ioannina
Other Study IDs: 234
Record Dates: First submitted 2019-02-20; First posted 2019-02-27 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2020-11

CONDITIONS: Dyslipidemias; Children, Only; Endothelial Dysfunction; Renal Dysfunction; Hypercholesteremia in Children
MeSH Terms: conditions — Dyslipidemias; Renal Insufficiency

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Serum
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Dyslipidemia group: Children and adolescents with dyslipidemia
- Control group: Children and adolescents without dyslipidemia

SUMMARY:
The aim of the study is to assess if abnormal lipid levels in childhood could cause early damage of the inner layer of the vessels, the endothelium. Dysfunction of the endothelium is the first event in the development of atherosclerosis, is present at all stages of atherosclerosis and is potentially reversible in childhood. It has been suggested that dyslipidemia, via its detrimental effects on endothelium, could impair renal function. This study will assess the dysfunction of the kidneys in children with dyslipidemia.

DETAILED DESCRIPTION:
In children recruited in the study, family history of dyslipidemia or premature cardiovascular disease will be recorded. Furthermore, anthropometric and clinical characteristics will be noted and lipid measurements will be obtained at recruitment after a fasting period.

The investigators will test in children the flow-mediated dilation (FMD) which assesses the vasodilation due to the production of nitric oxide from the endothelium in response to occlusion-induced hyperaemia of the branchial artery and the carotid intima-media thickness (cIMT). These non-invasive ultrasound indices detect early vascular damage.

Renal function will be assessed in children with dyslipidemia by a new marker in serum, cystatin C, which is more accurate and reliable than creatinine. Also, creatinine serum levels and estimated glomerular filtration rate (eGFR) will be evaluated. Additionally, total protein, albumin, electrolyte and β2-microglobulin excretion in urine will be measured.

ELIGIBILITY:
Inclusion Criteria:

* Children and adolescents aged 7 to 17 years
* Dyslipidemia (serum levels of LDL-cholesterol ≥95th percentile or serum levels of triglycerides ≥95th percentile or serum levels of HDL-cholesterol ≤5th percentile for age and sex)

Exclusion Criteria:

* History of renal disease
* Dyslipidemia caused by nephrotic syndrome or chronic kidney disease
* Chronic use of medication
* Acute or chronic inflammatory process

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The group of children with dyslipidemia will be selected from children referred to the Outpatient Lipid Clinic for Children and Adolescents and to the Pediatric Nephrology Department of the University Hospital of Ioannina. These are centers of excellence for assessing children with dyslipidemia and renal function in Northwestern Greece.
  The referrals are due to abnormal lipid levels in routine blood samples or family history of dyslipidemia and/or family history of premature cardiovascular disease.
  The group of controls will be selected from children attending the Outpatient Pediatric Clinic of University Hospital of Ioannina for follow-up of headache, heart murmur, constipation and loss of consciousness.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2017-04-03 (Actual); Primary Completion 2020-04-03 (Actual); Study Completion 2020-04-03 (Actual)

PRIMARY OUTCOMES:
Flow-mediated dilation of the branchial artery | At subject enrollment
  Non-invasive ultrasound assessment of endothelial function.
Carotid intima-media thickness | At subject enrollment
  Non-invasive ultrasound assessment of early vascular disease.
Measurement of cystatin C in serum | At subject enrollment
  Cystatin C is a marker for assessing renal function

SECONDARY OUTCOMES:
Number of participants with abnormal levels of lipoprotein a. | At subject enrollment
Levels of β2-microglobulin in urine | At subject enrollment
  Assessment of tubular function of the kidneys.
Serum creatinine levels | At subject enrollment
  Assessment of renal function
Assessment of eGFR | At subject enrollment

CONTACTS AND LOCATIONS:
Locations (1):
- University of Ioannina, Ioannina, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kosmeri C, Siomou E, Vlahos AP, Milionis H. Review shows that lipid disorders are associated with endothelial but not renal dysfunction in children. Acta Paediatr. 2019 Jan;108(1):19-27. doi: 10.1111/apa.14529. Epub 2018 Aug 22. PMID 30066344
- [Derived] Kosmeri C, Milionis H, Vlahos AP, Benekos T, Bairaktari E, Cholevas V, Siomou E. The impact of dyslipidemia on early markers of endothelial and renal dysfunction in children. J Clin Lipidol. 2021 Mar-Apr;15(2):292-300. doi: 10.1016/j.jacl.2020.12.003. Epub 2020 Dec 11. PMID 33478934